CLINICAL TRIAL: NCT02201160
Title: Impact of n-3 Fatty Acid Supplementation on the Metabolic Abnormalities in Children With NAFLD
Brief Title: Potential Role of n-3 Fatty Acids in the Treatment of NAFLD in Pediatric Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Justine's Hospital (Other)
Collaborators: Nutrisanté Canada (Unknown)
Responsible Party: Principal Investigator, Emile Levy, Full professor and researcher, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NAFLD-2188
Record Dates: First submitted 2014-07-18; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Non Alcoholic Fatty Liver Disease (NAFLD)
Keywords: NAFLD; Fatty acid composition; Omega 3 supplementation; Metabolism
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- omega 3 (Active Comparator): The subjects will take 4 capsules/day during 6 months. Each capsule of the active n-3 PUFA supplement contained 500 mg of fish oil (each capsule provides 300 mg of n-3 PUFA (EPA+DHA) with 3.75 U vitamin E to prevent peroxidation).
  Interventions: Dietary Supplement: omega 3
- Sun Flower (Placebo Comparator): The subjects will take 4 capsules/day during 6 months. The placebo capsule contained 500 mg of sunflower oil with 3.75 U vitamin E.
  Interventions: Dietary Supplement: omega 3

INTERVENTIONS:
Dietary Supplement: omega 3 — Two groups from our cohort will be supplemented either with omega-3 PUFA or placebo during 3 months. Each subject will take 4 capsules/d. after 3 months, the subjects under omega-3 will continue for another 3 months and the group under placebo will take omega-3 PUFA during another 3 months.

SUMMARY:
Nonalcoholic hepatic steatosis (NASH) is defined as the amount greater than 5% of the total liver volume fat. Commonly known as NASH, it includes 4 stages histological ranging from the mere presence of fat to the existence of fibrosis and degeneration of hepatocytes, and finally a progression to cirrhosis, sometimes accompanied by complications of hepatocellular carcinoma. It is a common condition associated with a combination of disorders, namely obesity, insulin resistance and type 2 diabetes. The link with the metabolic syndrome (MetS) was mainly studied in the adult population and very little in the paediatric population, while 15 and 25% of obese children are affectés. The severity of histological disease appears to be associated with the degree of obesity in children and particularly in the MetS. in addition, epidemiological data indicate that the incidence of this disease is increasing in children and positioning as the first NASH liver disease in North America. the revelation of the factors associated with the occurrence of NASH is a first necessary step to understanding this disorder worrying for the future of children and adolescents. In addition, clarification of the mechanisms responsible for its development is essential if the investigators want to consider targeted and effective treatments to slow the rat race of NASH, which stands out as the supreme chronic liver accompanying the obesity and MetS. Finally, in view of growth and puberty of children, it would be extremely beneficial to find nutritional avenues that would avoid the side effects of chemical agents.

DETAILED DESCRIPTION:
The aims of the investigators studies are to determine the plasma FA composition and to assess changes in the latter in response to n-3 supplementation in French-Canadian youth since (i) none of the available pharmacological agents could be recommended for treatment of children with NAFLD; (ii) n-3 PUFA are quite safe diet supplements that showed efficacy in the prevention and therapy of cardiovascular diseases, dyslipidemia and metabolic syndrome; (iii) loss of n-3 PUFA dietary intake was found in pediatric NAFLD and (iii) no attention has been given to French-Canadian population, which is primarily and historically located in the province of Quebec, has the highest prevalence worldwide of lipoprotein lipase deficiency, includes a large pool of individuals at risk for atherosclerosis and other lipid-related diseases, and exhibits a founder effect among the 8,000 ancestors of present-day French-Canadians, who have had relatively little cross-breeding with individuals from other national origin groups.

Subjects The present randomized clinical trial was performed on 30 NAFLD children followed as outpatients at the Gastroenterology/Hepatology and Nutrition clinic of MCHU Ste-Justine and the Gastroenterology division of the Montreal Children's Hospital, Montreal.

The children have between 8 years and 18 years of age, with obesity and a diagnostic of NAFLD based on the results of a clinical evaluation, liver echography, and magnetic resonance imaging-proton density fat fraction.

Inclusion and exclusion criteria The children are eligible for the study if they are boys (according to the literature review on NAFLD prevalence), with a body weight ≥ 95th percentile (based on the CDC Chart), aged <18 years, have a diffusely hyperechogenic liver at ultrasonography (consistent with NAFLD diagnostic), and have normal or high transaminases (> 2N). Moreover, the exclusion criteria is based on subjects having pin or cochlear implants may affect the magnetic resonance imaging examination; subjects who consumed natural medicine products have an increased risk of haemorrhage, and those in whom a surgical procedure was planned, and the child who founded to consume fish, flaxseed oil and foods enriched with n-3 PUFA (eggs, or milk containing n-3 PUFA supplements), probiotics, vitamin E or use of drugs known to induce fatty liver during the study.

Study design The present study is a 6-month, double-blind, one-way, crossover randomized study. The treatment consisting of n-3 PUFA supplement (NutriSanté Inc./Ponroy, Canada), administered in two phases, each of 3-month duration. In the first phase, an NAFLD group will receive an active n-3 PUFA supplement and another will receive equivalent quantities of sunflower oil as a placebo. During the second phase (after the first 3 months), all NAFLD subjects will receive an active n-3 PUFA. The study is approved by the Clinical Research Ethics Committee of MUCH Ste-Justine (Montreal, Quebec. Informed consent was obtained from all subjects before starting experimental procedures, and the study followed the Helsinki guidelines.

Dosing The dose supplementation considered for this study is 2.0 g of fish oil per day, providing a total of 1.2 g of n-3 PUFA. This dose is chosen according to official recommendations, based on our previous studies and pediatric clinical trials. Compliance to the study treatment will be evaluated by pill count at every visit, review of medication records, and direct interview of patients by the physician.

ELIGIBILITY:
Inclusion Criteria:

* boys (according to the literature review on NAFLD prevalence)
* body weight ≥ 95th percentile (based on the CDC Chart)
* aged <18 years
* have a diffusely hyperechogenic liver at ultrasonography (consistent with NAFLD diagnostic)
* have normal or high transaminases (> 2N).

Exclusion Criteria:

* Subjects with pin or cochlear implants
* Subjects who consumed natural medicine products
* Those in whom a surgical procedure was planned
* the child who were found to consume fish, flaxseed oil and foods enriched with n-3 PUFA (eggs, or milk containing n-3 PUFA supplements), probiotics, vitamin E or use of drugs known to induce fatty liver during the study.

Ages: 8 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of omega 3 PUFA supplementation in NAFLD subjects compared to placebos | 24 weeks
  Two groups from our cohort will be double blind supplemented either with n-3 PUFA or sun flower (as a placebo).
  The specific primary outcome is to assess the activities of hepatic plasma transaminase enzymes (ALT/AST/GGT) in the omega 3 group and to determine their decrease to the normal range.

SECONDARY OUTCOMES:
A composite mesures regarding the improvement of metabolic profile of NAFLD patients | 24 weeks
  To determine
  * the decrease in obesity (body mass index)
  * insulin resistance (HOMA-IR)
  * Adipose tissue lowering (DEXA)
  * Oxidative stress (Malondialdehyde biomarker, oxLDL) Inflammation (TNFalpha, IL-6, leptin and resistine)
  * Plasma lipids (triglycerides, total cholesterol, LDL and HDL cholesterol)

OTHER OUTCOMES:
Short term versus long-term treatment comparison | 12 weeks vs. 24 weeks
  To compare the effectiveness of omega 3 PUFA between 12- and 24-weeks by a composite measures in terms of percent decrease in the
  * transaminases (ALT/AST/GGT)
  * body weight (BMI)
  * Insulin resistance (HOMA-IR)
  * Oxidative stress (malondialdehyde marker)
  * Inflammation (TNF-alpha, interleukin-6, leptin and resistin)
  * Lipids (triglycerides, cholesterol, LDL-cholesterol, HDL-cholesterol)
  * changes in adipose tissue (DEXA)

CONTACTS AND LOCATIONS:
Overall Officials: Emile Levy, Professor, Principal Investigator — Research Centre, CHU STe-Justine
Locations (1):
- CHU Ste-Justine, Montreal, Quebec, Canada

REFERENCES:
- [Background] Belanger SA, Vanasse M, Spahis S, Sylvestre MP, Lippe S, L'heureux F, Ghadirian P, Vanasse CM, Levy E. Omega-3 fatty acid treatment of children with attention-deficit hyperactivity disorder: A randomized, double-blind, placebo-controlled study. Paediatr Child Health. 2009 Feb;14(2):89-98. doi: 10.1093/pch/14.2.89. PMID 19436468
- [Derived] Spahis S, Alvarez F, Ahmed N, Dubois J, Jalbout R, Paganelli M, Grzywacz K, Delvin E, Peretti N, Levy E. Non-alcoholic fatty liver disease severity and metabolic complications in obese children: impact of omega-3 fatty acids. J Nutr Biochem. 2018 Aug;58:28-36. doi: 10.1016/j.jnutbio.2018.03.025. Epub 2018 Apr 10. PMID 29864682